CLINICAL TRIAL: NCT02470039
Title: An 8-week Randomised, Double-blind, Parallel, Multiple Dose Trial Comparing NNC0123-0000-0338 in a Tablet Formulation and Insulin Glargine in Subjects With Type 2 Diabetes Currently Treated With Oral Antidiabetic Therapy
Brief Title: Trial to Compare NNC0123-0000-0338 in a Tablet Formulation and Insulin Glargine in Subjects With Type 2 Diabetes Currently Treated With Oral Antidiabetic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1953-4163; 2014-002716-16 (EudraCT Number); U1111-1158-3620 (Other: WHO)
Record Dates: First submitted 2015-05-29; First posted 2015-06-12 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral insulin 338 and subcutaneous placebo (Experimental)
  Interventions: Drug: insulin 338 (GIPET I); Drug: placebo
- Subcutaneous insulin glargine and oral placebo (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: placebo

INTERVENTIONS:
Drug: insulin 338 (GIPET I) — Oral administered once daily in combination with metformin with or without DPP-4 inhibitor
  Arms: Oral insulin 338 and subcutaneous placebo
Drug: insulin glargine — Injected s.c./subcutaneously (under the skin) once daily in combination with metformin with or without DPP-4 inhibitor
  Arms: Subcutaneous insulin glargine and oral placebo
Drug: placebo — Administered once daily

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare NNC0123-0000-0338 (insulin-338) in a tablet formulation and insulin glargine in combination with metformin with or without DPP-4 inhibitor in subjects with type 2 diabetes currently treated with oral antidiabetic therapy

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-70 years (both inclusive) at the time of signing informed consent
* Body mass index of 25.0-40.0 kg/m^2 (both inclusive)
* Subject diagnosed (clinically) with type 2 diabetes mellitus for at least 180 days prior to the day of screening
* Insulin naïve subject; however, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes

Exclusion Criteria:

* Known or suspected hypersensitivity to the trial products or related products
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma glucose (FPG) | Week 0, Week 8

SECONDARY OUTCOMES:
Change from baseline in 10-points plasma glucose profile | Week 0, Week 8
Number of treatment emergent hypoglycaemic episodes | From start of treatment until Visit 14 (Day 68)
area under the serum insulin concentration-time curve | During one dosing interval (0 to 24 hours) at steady state (Day 56)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

REFERENCES:
- [Result] Halberg IB, Lyby K, Wassermann K, Heise T, Zijlstra E, Plum-Morschel L. Efficacy and safety of oral basal insulin versus subcutaneous insulin glargine in type 2 diabetes: a randomised, double-blind, phase 2 trial. Lancet Diabetes Endocrinol. 2019 Mar;7(3):179-188. doi: 10.1016/S2213-8587(18)30372-3. Epub 2019 Jan 21. PMID 30679095
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com